CLINICAL TRIAL: NCT02321410
Title: Plaque Neovascularization Assessment by Contrast Ultrasounds and Plaque Magnetic Resonance: "in Vivo" Comparison in Human Carotid Atherosclerosis
Brief Title: "In Vivo" Comparison in Human Carotid Atherosclerosis: Plaque Neovascularization
Acronym: PLAVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Giovanni Bellinzona (Other)
Responsible Party: Principal Investigator, Professor Augusto Gallino, Professor MD, Ospedale San Giovanni Bellinzona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE 2674
Record Dates: First submitted 2014-11-26; First posted 2014-12-22 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Carotid Artery Disease; Plaque Neovascularization
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging of carotid plaque (Other): Patient undergo contrast enhanced ultrasound of the carotid plaque and dynamic contrast-enhanced carotid plaque MRI
  Interventions: Other: Contrast enhanced ultrasound of the carotid plaque; Other: Dynamic contrast-enhanced carotid plaque MRI

INTERVENTIONS:
Other: Contrast enhanced ultrasound of the carotid plaque — visual grading of neovessel
Other: Dynamic contrast-enhanced carotid plaque MRI — quantitative analysis of gadolinium enchantment in a region of interest

SUMMARY:
Atherosclerosis may initiate early in life and takes years to progress. This contrasts to the abrupt coronary or cerebrovascular events occurring following the transition from a stable to an unstable atherosclerotic plaque. The causes of this discontinuity of the disease are complex and probably multiple. There is increasing evidence that, besides inflammation, neovascularisation of atherosclerotic plaques and intra-plaque hemorrhages play an important role in plaque instability ending-up frequently in acute thrombotic occlusion or distal embolisation of athero-thrombotic material associated with heart attack or stroke. Contrast-enhanced Ultrasound, is a bed-side non-invasive technique, which allows to enhance microvascular structures and to visualize the adventitia and intraplaque vascularization. Dynamic contrast-enhanced plaque MRI (DCE-MRI) which has also been evaluated for in vivo detection and quantification of plaque neovascularity. Together with the presence of a large lipid-rich core, thin fibrous cap, positive remodeling and active inflammatory infiltrate, plaque neovascularisation is considered a valid marker of high-risk (or vulnerable) plaque as demonstrated in histopathological studies using microvessel density.

Aim of the study is to assess and validate the value of contrast enhanced ultrasound (CEUS), a bed-side technique, in detecting plaque neovascularisation and compare it with the quantitative assessment by DCE-MRI in carotis atherosclerosis.

A group of 30 patients with asymptomatic carotid atherosclerosis (> 50% stenosis on Doppler ultrasound) will undergo Carotid Duplex ultrasounds and CEUS. High-resolution plaque MRI and DCE-MRI will be performed in the same patients and will be analyzed by two separate operators blinded to the results of the CEUS in order to detect the efficacy of CEUS when compared with in vivo DCE-MRI, as the standard of reference.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic 50-70% carotid artery stenosis on Doppler ultrasound
* Asymptomatic >70% carotid artery stenosis on Doppler ultrasound (no surgical indication)
* Signed informed consent

Exclusion Criteria:

* Non atherosclerotic occlusive disease
* Prior carotid endarterectomy on the site of the index carotid artery
* Contraindications for MRI and CE MRI (history of hypersensitivity to gadolinium salt, pacemaker or vascular clip implantation, implantation of any metallic device, severe claustrophobic reactions)
* Contraindications to CEUS (hypersensitivity to Sonovue compounds, acute coronary syndromes, acute heart failure, heart failure in NYHA class III or IV, severe arrhythmias, known right-to-left cardiac shunt, severe pulmonary hypertension, uncontrolled arterial hypertension, acute distress respiratory syndrome)
* Short-term life-threatening pathology (life expectancy < 6 months)
* Physically unable to participate in the study
* Compliance not guaranteed
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Plaque neovascularization grading and quantification (assessment by DCE-MRI) | Baseline
  Contrast enhanced ultrasound plaque neovascularization grading , correlated to plaque neovascularization quantitative assessment by DCE-MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Gallino, Prof. MD, Principal Investigator — Ospedale Regionale di Bellinzona e Valli - Ospedale San Giovanni Bellinzona; Mattia Cattaneo, MD, Study Chair — Ospedale Regionale di Bellinzona e Valli - Ospedale San Giovanni Bellinzona
Locations (1):
- Ospedale Regionale di Bellinzona e Valli - Ospedale San Giovanni Bellinzona, Bellinzona, Canton Ticino, Switzerland

REFERENCES:
- [Result] Cattaneo M, Staub D, Porretta AP, Gallino JM, Santini P, Limoni C, Wyttenbach R, Gallino A. Data on consistency among different methods to assess atherosclerotic plaque echogenicity on standard ultrasound and intraplaque neovascularization on contrast-enhanced ultrasound imaging in human carotid artery. Data Brief. 2016 Oct 3;9:563-567. doi: 10.1016/j.dib.2016.09.041. eCollection 2016 Dec. PMID 27752526
- [Result] Cattaneo M, Staub D, Porretta AP, Gallino JM, Santini P, Limoni C, Wyttenbach R, Gallino A. Contrast-enhanced ultrasound imaging of intraplaque neovascularization and its correlation to plaque echogenicity in human carotid arteries atherosclerosis. Int J Cardiol. 2016 Nov 15;223:917-922. doi: 10.1016/j.ijcard.2016.08.261. Epub 2016 Aug 16. PMID 27597156
- [Derived] Cattaneo M, Sun J, Staub D, Xu D, Gallino JM, Santini P, Porretta AP, Yuan C, Balu N, Arnold M, Froio A, Limoni C, Wyttenbach R, Gallino A. Imaging of Carotid Plaque Neovascularization by Contrast-Enhanced Ultrasound and Dynamic Contrast-Enhanced Magnetic Resonance Imaging. Cerebrovasc Dis. 2019;48(3-6):140-148. doi: 10.1159/000504042. Epub 2019 Oct 29. PMID 31661690